CLINICAL TRIAL: NCT05643534
Title: A 12-Week, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Assess the Safety and Efficacy of Tenapanor for the Treatment of Irritable Bowel Syndrome With Constipation (IBS-C) in Pediatric Patients 12 to Less Than 18 Years Old
Brief Title: Study to Assess Safety and Efficacy of Tenapanor for Treatment of IBS-C in Pediatric Patients 12 to Less Than 18 Years
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ardelyx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TEN-01-304
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Irritable Bowel Syndrome With Constipation (IBS-C)
Keywords: IBS-C
MeSH Terms: interventions — tenapanor; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tenpanor 50 mg BID (Experimental): Patients will be randomized to receive 50 mg tenapanor twice daily
  Interventions: Drug: Tenapanor 50 MG
- Tenpanor 25 mg BID (Experimental): Patients will be randomized to receive 25 mg tenapanor twice daily
  Interventions: Drug: Tenapanor 25 mg bid
- Placebo Comparator (Placebo Comparator): Patients will be randomized to receive matching placebo twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tenapanor 50 MG — Participants will receive tenapanor 50 mg BID (total of 100 mg daily)
  Arms: Tenpanor 50 mg BID
Drug: Tenapanor 25 mg bid — Participants will receive tenapanor 25 mg BID (total of 50 mg daily)
  Arms: Tenpanor 25 mg BID
Drug: Placebo — Participants will be randomized to receive matching placebo
  Arms: Placebo Comparator

SUMMARY:
This is a randomized, double-blind, placebo-controlled study to assess the efficacy, safety and tolerability of tenapanor (25 mg and 50 mg) in pediatric patients (≥12 and <18 years old) with IBS-C when administered twice daily (BID) for 12 consecutive weeks.

DETAILED DESCRIPTION:
This study consists of 2-week screening period followed by 12 week randomized treatment period (RTP) and a 2-week treatment-free Follow-Up period (only for patients who will not enter the 40-week Long Term Safety Extension Study [TEN-01-306]). At the beginning of the 2-week Screening period, patients who provide written assent will be fully assessed for eligibility into the study and will be asked to self-report daily information about the status of their IBS symptoms via an electronic diary (eDiary) device. Patient compliance with the eDiary will be monitored actively by the site staff and will be reviewed to determine eligibility at the end of screening. Eligible patients will be randomized to receive one of the study medications: tenapanor 25 mg BID, tenapanor 50 mg BID, or placebo.

During the 12-week double-blind RTP, patients will continue recording daily assessments via the eDiary system as instructed and compliance with eDiary entries will be monitored on an ongoing basis. Patients will return for study visit every two or four weeks (Visits 3-6) and will undergo safety assessments at these visits.

Patients who do not enter the 40-week Long Term Safety Extension Study [TEN-01-306] including those who complete the RTP but do not enter study TEN-01-306 and those who prematurely discontinue from the RTP, a Follow-Up Visit will be scheduled approximately 2 weeks after the completion of the RTP (Visit 6) or the Early Termination Visit at which safety assessments will be performed

ELIGIBILITY:
Inclusion Criteria:

* ≥12 and <18 years old
* Patient weighs ≥18 kg at the time the patient provides written assent
* Females of child-bearing potential must have negative pregnancy test at Visit 1 (serum) and Visit 2 (urine) and confirm the use of appropriate contraception (including abstinence).
* Patient meets the Rome IV criteria for child/adolescent diagnosis of IBS-C
* Patient is willing to discontinue any laxatives used in favor of the protocol-permitted rescue medicine (which will only be allowed after 72 hours with no bowel movement)
* Patient meets the entry criteria assessed during the 2-week Screening period.
* Ability of both the patient and parent/guardian/LAR to communicate with the Investigator and to comply with the requirements of the entire study, including an understanding of the assessments in the eDiary and how to use the eDiary device
* Patient must provide written assent and the parent/guardian/LAR must provide written informed consent before the initiation of any study-specific procedures

Exclusion Criteria:

* Functional diarrhea as defined by Rome IV child/adolescent criteria
* IBS with diarrhea (IBS-D), mixed IBS (IBS-M), or unsubtyped IBS as defined by Rome IV child/adolescent criteria
* History of non-retentive fecal incontinence.
* Required manual disimpaction any time prior to randomization (after consent);
* Has both unexplained and clinically significant alarm symptoms (lower gastrointestinal [GI] bleeding [rectal bleeding or heme-positive stool], iron-deficiency anemia, or any unexplained anemia, or weight loss) and systemic signs of infection or colitis, or any neoplastic process
* Patient has any of the following conditions:

  * Celiac disease, or positive serological test for celiac disease
  * Cystic fibrosis
  * Hypothyroidism that is untreated or treated with thyroid hormone
  * Down's syndrome or any other chromosomal disorder
  * Active anal fissure
  * Anatomic malformations (eg, imperforate anus)
  * Intestinal nerve or muscle disorders (eg, Hirschprung disease)
  * Neuropathic conditions (eg, spinal cord abnormalities)
  * Lead toxicity, hypercalcemia
  * Neurodevelopmental disabilities producing a cognitive delay that precludes comprehension and completion of the daily eDiary (Electronic handheld device)
  * Inflammatory bowel disease
  * Childhood functional abdominal pain syndrome
  * Childhood functional abdominal pain;
  * Poorly treated or poorly controlled psychiatric disorders that might influence his or her ability to participate in the study;
  * Lactose intolerance that is associated with abdominal pain or discomfort
  * History of cancer other than treated basal cell carcinoma of the skin; (Note: Patients with a history of cancer are allowed provided that the malignancy has been in a complete remission for at least 5 years before the Randomization Visit.)
  * History of diabetic neuropathy.
* Use of medications that are known to affect stool consistency (Prohibited Medications), including fiber supplements, anti-diarrheals, cathartics, antacids, opiates, prokinetic drugs, laxatives, enemas, antibiotics during the Screening period; unless specified as rescue medication, and used accordingly as directed by the Investigator.
* Patient has had surgery that meets any of the following criteria:

  * Bariatric surgery for treatment of obesity, or surgery to remove a segment of the GI tract at any time before the Screening Visit;
  * Surgery of the abdomen, pelvis, or retroperitoneal structures during the 6 months before the Screening Visit;
  * An appendectomy or cholecystectomy during the 60 days before the Screening Visit;
  * Other major surgery during the 30 days before the Screening Visit
* History of alcohol or substance abuse
* Participation in other clinical trials within 1 month prior to Screening
* Patient and/or parent/guardian/LAR is involved in the conduct and/or administration of this trial as an investigator, sub-investigator, trial coordinator, or other staff member, or the patient is a first-degree family member, significant other, or relative residing with one of the above persons involved in the trial
* If, in the opinion of the Investigator, the patient is unable or unwilling to fulfill the requirements of the protocol or has a condition, which would render the results uninterpretable

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
6/12-week APS (abdominal pain and SBM) +2 response | 12 weeks
  6/12-week APS (abdominal pain and SBM (spontaneous bowel movement)) +2 response, defined as achieving the weekly APS +2 response criteria (i.e., achieving both weekly SBM +2 response and weekly abdominal pain response during the same week) for ≥6 out of the 12 weeks of the RTP.
  * The weekly SBM +2 response is defined as having an increase of ≥2 from baseline in the average weekly SBM frequency for a given week
  * The weekly abdominal pain response is defined as having ≥30% reduction from baseline in the average weekly abdominal pain score for a given week

SECONDARY OUTCOMES:
6/12-week SBM +2 response | 12 weeks
  6/12-week SBM +2 response: defined as achieving the weekly SBM +2 response for ≥6 out of the 12 weeks of the RTP
6/12-week abdominal pain response | 12 weeks
  6/12-week abdominal pain response: defined as achieving the weekly abdominal pain response for ≥6 out of the 12 weeks of the RTP
Change from baseline in average weekly SBM frequency | 12 weeks
  Change from baseline in average weekly SBM frequency
Change from baseline in average weekly stool consistency score | 12 weeks
  Change from baseline in average weekly stool consistency score
Change from baseline in average weekly abdominal pain score | 12 weeks
  Change from baseline in average weekly abdominal pain score
Overall use of rescue medication | 12 weeks
  Overall use of rescue medication

CONTACTS AND LOCATIONS:
Overall Officials: Susan Edelstein, PhD, Study Director — Ardelyx
Locations (41):
- United States (41):
  - G & L Research, LLC, Foley, Alabama
  - Eclipse Clinical Research, Tucson, Arizona
  - Advanced Research Center, Inc., Anaheim, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Prohealth Research Center, Doral, Florida
  - I.H.S. Health, LLC, Kissimmee, Florida
  - Waterway Research & Associates Corp, Miami, Florida
  - Valencia Medical and Research Center, Miami, Florida
  - Orlando Health, Inc.- APH Center for Digestive Health and Nutrition, Orlando, Florida
  - Florida Pharmaceutical Research and Associates, Inc., South Miami, Florida
  - Clinical Research Institute, Stockbridge, Georgia
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Riley Children's Health IUH, Indianapolis, Indiana
  - Maine Health, Portland, Maine
  - Boston Children's Hospital, Boston, Massachusetts
  - Mankato Clinic/ Javara Research Ltd, Mankato, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Boys Town National Research Hospital, Boys Town, Nebraska
  - Med Clinical Research Partners, LLC, Irvington, New Jersey
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - SUNY Downstate Medical Center, Brooklyn, New York
  - University of Rochester, Rochester, New York
  - Advantage Clinical Trials, The Bronx, New York
  - Atrium Health, Charlotte, North Carolina
  - Duke University School of Medicine, Durham, North Carolina
  - M3 Wake Research, Inc, Raleigh, North Carolina
  - Wilmington Health, Wilmington, North Carolina
  - Frontier Clinical Research, LLC, Scottdale, Pennsylvania
  - Frontier Clinical Research, LLC, Smithfield, Pennsylvania
  - Velocity Clinical Research, Providence, East Greenwich, Rhode Island
  - Prisma Health Children's Hospital, Greenville, South Carolina
  - Advance Clinical Trial PLLC, Abilene, Texas
  - Maspons Pediatric Gastro, El Paso, Texas
  - Proactive El Paso, LLC, El Paso, Texas
  - Texas Digestive Specialists, Harlingen, Texas
  - AIM Trials, LLC, Plano, Texas
  - Sun Research Institute, San Antonio, Texas
  - Pioneer Research Solutions Inc, Sugar Land, Texas
  - ClinPoint Trials, Waxahachie, Texas
  - University Physicians and Surgeons, Inc., Huntington, West Virginia
  - Frontier Clinical Research, Kingwood, West Virginia

IPD SHARING:
Plan to Share IPD: No